CLINICAL TRIAL: NCT05284214
Title: Sargramostim Safety and Tolerability With Standard Of Care Ipilimumab Containing Therapy in Patients With Solid Tumors
Brief Title: Sargramostim With Ipilimumab Containing Therapy in Patients With Solid Tumors
Acronym: SALIENT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not commence.
Sponsor: Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTX-001-004
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor; Solid Tumor, Adult
MeSH Terms: interventions — sargramostim; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sargramostim daily: 14 of 21 days (Experimental): Sargramostim administered by subcutaneous (SC) injection for 14 consecutive days every 3 weeks, for up to 12 weeks, given in combination with an ipilimumab-containing regimen.
  Interventions: Biological: Sargramostim; Biological: Ipilimumab-containing therapy
- Sargramostim daily: 5 of 7 days (Experimental): Sargramostim given by SC injection for 5 consecutive days every week, for up to 12 weeks, given in combination with an ipilimumab-containing regimen for a total of 12 weeks.
  Interventions: Biological: Sargramostim; Biological: Ipilimumab-containing therapy

INTERVENTIONS:
Biological: Sargramostim — Sargramostim for injection
  Other Names: Leukine®
Biological: Ipilimumab-containing therapy — Treatment for cancer containing ipilimumab at either 1 mg/kg or 3 mg/kg, intravenously..
  Other Names: Yervoy®

SUMMARY:
This open label, randomized study will evaluate safety and tolerability of sargramostim when combined with an ipilimumab-containing regimen received as part of standard of care therapy. The study will evaluate 2 sargramostim administration schedules. Patients will be randomized 1:1 to the sargramostim administration schedules and stratified based on planned dose of ipilimumab (1 mg/kg, 3 mg/kg).

Sargramostim will be administered for the first 12 weeks following the assigned treatment schedule or until disease progression, intolerable toxicity, consent withdrawal, pregnancy, or death, whichever comes first. Checkpoint inhibitor therapy will be administered in accordance with institutional standard of care guidelines, at the Investigator's discretion.

Patients will be followed up for to 24 weeks following end of sargramostim treatment for safety, efficacy, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with solid tumors that will start an ipilimumab-containing therapy (with or without anti-PD-1, such as nivolumab) as part of standard of care in approved ipilimumab indication
* Recovery from any toxicities related to prior therapies
* Ability and willingness to self-administer or have a caregiver administer a SC injection of sargramostim
* Women of child-bearing potential willing to use birth control

Exclusion Criteria:

* Recent radiation therapy for cancer that has spread to bones or to the brain
* History of a severe reaction to prior immune checkpoint inhibitors
* Pleural or pericardial effusion, or history of recurrent pleural or pericardial effusion.
* Heart rhythm with symptoms within the last 12 months
* Known or suspected intolerance or hypersensitivity to sargramostim or any product component or diluent
* Use drugs that can suppress the immune system
* Women who are pregnant or breastfeeding
* Live virus vaccine within 28 days prior to study treatment and for 4 weeks after study treatment.
* Have other active cancers
* Participation in another clinical trial
* Any other medical condition or laboratory abnormality that would put patient at risk or confound interpretation of trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The number of participants with severe, life-threatening or fatal adverse events | Up to 36 weeks

SECONDARY OUTCOMES:
Number of participants who develop colon inflammation (colitis) | Up to 36 weeks
Number of participants who develop pneumonitis (lung inflammation) | Up to 36 weeks
Number of participants who discontinue sargramostim due to a treatment related adverse event | Up to 12 weeks
Number of missed doses | Up to 12 weeks
Number of participants requiring dose modifications | Up to 12 weeks
Change from baseline in Treatment Assessment Questionnaire | Daily up to 12 weeks.
Number of participants who develop anti-drug antibodies against sargramostim | Day 1, Week 4, Week 13, Week 17 and Week 36
Overall response rate | Up to Week 36
  The number of participants who have a complete response or partial response to treatment using Investigator-assessed efficacy evaluation by immune-related (i)Response Evaluation Criteria in Solid Tumors (iRECIST):
Disease control rate | Up to Week 36
  The number of participants who have a complete response, partial response, or stable disease response to treatment using Investigator-assessed efficacy evaluation by iRECIST:
Progression-free survival | Up to 36 weeks
  The time from randomization until disease progression or death from any cause
Overall survival | Up to 36 weeks
  The time from randomization until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Garner, Study Director — Partner Therapeutics, Inc.
Locations (1):
- Partner Therapeutics - No Currently Active Sites, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided